CLINICAL TRIAL: NCT06706635
Title: Impact of Enhanced Information Provision by Using a Mobile App on Subjective Information Level As the Basis for Shared-decision Making and Patient-reported Outcome Measures (PROMs) in Patients with Aortic Stenosis
Brief Title: Impact of Enhanced Information on Subjective Information Level and PROMs in Patients with Aortic Stenosis
Acronym: TAVI-SDM-APP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HDZ-KA_023_TR
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Aortic Stenosis Disease
Keywords: aortic stenosis; mobile app
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full access to a mobile App (Experimental): Study patients will receive full access to a mobile App
  Interventions: Device: Application of App
- Restricted access to a mobile App (Other): Study patients will receive restricted access to a mobile App
  Interventions: Device: Application of App

INTERVENTIONS:
Device: Application of App — Full Access to Mobile App

SUMMARY:
The aim of this trial is to evaluate if an enhanced information by using a mobile App can increase subjective information level in patients with severe aortic stenosis and may therefore improve patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* severe aortic valve stenosis
* planned aortic valve replacement (TAVI)
* Patient is willing and able to complete the surveys in German language
* Written informed consent by the trial subject

Exclusion Criteria:

- Language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Subjective information level (EORTC QOL-INFO 25 questionnaire) | From enrollment to the end of FU at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for General and Interventional Cardiology/Angiology, Herz- und Diabeteszentrum NRW, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No